CLINICAL TRIAL: NCT03635346
Title: Medicinal Dependence and Chronic Pain: Addictive Evaluation in CETD
Acronym: DEMDOU
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: DEMDOU 2016.CE13
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-07

CONDITIONS: Opiate Dependence; Chronic Pain
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
prescription opioid misuse in chronic pain is a growing public health concern. few studies got interested in prevalence of misuse and of opiate use disorder in a population of patients with a non cancer chronic pain.

the investigators analyzed during 3 months opiate misuse and opiate ude disorder in a population of patients consulting a center specialized in pain management.

ELIGIBILITY:
Inclusion Criteria:

* patient with a non cancer chronic pain
* consulting a CETD center

Exclusion Criteria:

* non understanding of french

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: analysis of SUD criteria in a population with a chronic pain (non cancer) , consulting a center specialized in pain mangement
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2016-09-03 (Actual); Study Completion 2018-03-10 (Actual)

PRIMARY OUTCOMES:
DSM 5 criteria of SUD | Day 0 (at the inclusion)
  11 criteria of SUD

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France